CLINICAL TRIAL: NCT04167748
Title: GEnetic Testing in Elective Single Embryo Transfer in Women of Advanced Maternal Age
Brief Title: Preimplantation Genetic Testing in Women of Advanced Maternal Age
Acronym: GETSET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Genomic Prediction Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Genomic Prediction Inc 624
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation information will be handled by researcher coordinators only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGT-A transfer (Experimental): Transfer of single chromosomally normal (euploid) blastocyst after PGT-A
  Interventions: Procedure: Preimplantation genetic testing for aneuploidy (PGT-A)
- Untested blastocyst transfer (No Intervention): Transfer of single untested blastocyst based on embryo morphology criteria.

INTERVENTIONS:
Procedure: Preimplantation genetic testing for aneuploidy (PGT-A) — 24-chromosome screening for aneuploidy in the preimplantation embryo (blastocyst stage)
  Other Names: Preimplantation genetic screening (PGS)
  Arms: PGT-A transfer

SUMMARY:
The GETSET trial is a prospective randomized trial designed to evaluate the clinical outcomes of incorporating preimplantation genetic testing for aneuploidies (PGT-A) in elective single embryo transfer in women between 35 and 40 years of age.

DETAILED DESCRIPTION:
In this randomized controlled trial, a total of 240 patients divided evenly across the two participating IVF centers will be recruited. Patients will be randomized to a control and to a treatment group, each containing 120 participants.

Only patients with at least one evaluable blastocyst will be randomized. Patients will undergo ovarian hyper-stimulation, oocyte retrieval, fertilization and embryo culture per standard clinical protocol determined by IVF center.

In the control arm, patients will undergo a single frozen embryo transfer with an untested blastocyst with the best morphology. All other blastocysts with lower morphology will undergo trophectoderm biopsy on day 5, 6 or 7 and will be frozen. PGT-A results of the untransferred embryos will be revealed to the patient AFTER the outcome of the initial ET is known. If the initial transfer results in a non-conception cycle and additional euploid embryos are available for transfer, these cycles will be followed and their outcomes collected.

In the experimental arm, all embryos will be cultured to blastocyst and all viable blastocysts will undergo trophectoderm biopsy and PGT-A. PGT-A will be performed regardless of the number of blastocysts available. Patients will undergo frozen transfer of the single, best quality euploid blastocyst. If the initial transfer results in a non-conception cycle and additional embryos are available for transfer, these cycles will be followed and their outcomes collected until the embryo cohort is exhausted.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF of between 35 and 40 years of age at IVF cycle start
* Utilization of Intracytoplasmic Sperm Injection ICSI
* Utilization of ejaculated or testicular sperm
* Utilization of autologous or donor sperm
* All Controlled Ovarian Hyperstimulation (COH) protocols

Exclusion criteria:

* Patients with anovulatory Polycystic ovarian syndrome (PCOS)
* Utilization of donor oocytes
* Utilization of gestational carrier
* Recurrent Pregnancy Loss (RPL) defined as ≥ 3 consecutive miscarriages
* Recurrent Implantation Failure (RIF) defined as ≥ 3 more failed embryo transfers

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | Up to 18 months
  Number of patients who experience an ongoing pregnancy rate (>20 weeks of gestation) after their first embryo transfer

SECONDARY OUTCOMES:
Miscarriage rate | Up to 18 months
  Number of patients who experience a miscarriage after their first embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Nathan R Treff, PhD, Principal Investigator — Genomic Prediction
Locations (1):
- IVF Florida Reproductive Associates, Margate, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Electronic address: ASRM@asrm.org; Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. The use of preimplantation genetic testing for aneuploidy (PGT-A): a committee opinion. Fertil Steril. 2018 Mar;109(3):429-436. doi: 10.1016/j.fertnstert.2018.01.002. PMID 29566854
- [Background] Yang Z, Liu J, Collins GS, Salem SA, Liu X, Lyle SS, Peck AC, Sills ES, Salem RD. Selection of single blastocysts for fresh transfer via standard morphology assessment alone and with array CGH for good prognosis IVF patients: results from a randomized pilot study. Mol Cytogenet. 2012 May 2;5(1):24. doi: 10.1186/1755-8166-5-24. PMID 22551456
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996